CLINICAL TRIAL: NCT00199121
Title: An Open, Single-Arm, Multi-Center, Phase IV Pilot Study of Treatment of Antiretroviral Naive HIV-1 Infected Patients With Tenofovir Disoproxil Fumarate in Combination With Emtricitabine and Zidovudine
Brief Title: A Pilot Study of Triple NtRTI/NsRTI Therapy in Antiretroviral Naive HIV-1 Infected Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEAZE001
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-12-14 (Estimated); Status verified 2005-07

CONDITIONS: HIV
MeSH Terms: interventions — Zidovudine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Zidovudine (drug)

SUMMARY:
The purpose of this study is to evaluate the antiviral effect and durability of antiviral response (HIV-1 RNA PCR) and safety of a triple NtRTI/NsRTI therapy in antiretroviral naive patients. Patients will receive TDF plus FTC plus AZT for at least 48 weeks. Further objectives are to evaluate resistance pathways in failing patients treated with TDF/FTC/AZT and to evaluate a treatment strategy of sparing PIs and NNRTIs for later treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* HIV-1 positive
* antiretroviral treatment naive
* one CD4 count >200/ul within 14d prior to study drug administration
* one HIV-1 RNA PCR value >5000 and <100.000 cop/ml within 14d prior to study drug administration
* women of child bearing potential: negative serum pregnancy test within 14d of study
* ability to understand and provide written informed consent
* overall stable disease
* absence of clinical signs of lipodystrophy

Exclusion Criteria:

* alcohol or illicit drug use
* malabsorption syndrome or other gastrointestinal dysfunction
* clinically relevant pancreatitis/hepatitis within the last 6 months
* receiving other investigational drugs
* abnormal hemoglobin, neutrophil, platelet, AST/ALT, pancreatic amylase, creatinine clearance, total bilirubine levels within 14d prior to study
* pregnancy/breast-feeding
* radiation therapy or cytotoxic chemotherapeutic agents within 30d of study
* prior antiretroviral therapy at any time, investigational antiretrovirals trial at any time, HIV vaccine within 90d prior to study
* immunomodulating agents
* serious medical condition (diabetes, congestive heart failure, cardiomyopathy, or other cardiac dysfunction)
* active diagnosis of AIDS (except for cutaneous Kaposi Sarcoma)
* foscarnet therapy or other agent with documented activity against HIV-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Schlomo Staszewski, MD, Principal Investigator — Head of the HIV Treatment & Research Unit, Dept. of Internal Medicine II, Hospital of the Johann Wolfgang Goethe University Frankfurt/Main, Germany
Locations (1):
- HIV Treatment & Research Unit, Dept. of Internal Medicine II, Hospital of the Johann Wolfgang Goethe University Frankfurt/Main, Frankfurt am Main, Hesse, Germany